CLINICAL TRIAL: NCT00681122
Title: An International, Observational Study to Evaluate the Impact of Educational Material on the Compliance and Persistence Rates to Adjuvant Aromatase Inhibitor (AI) Medication for Postmenopausal Woman
Brief Title: CARIATIDE (Compliance of ARomatase Inhibitors AssessmenT In Daily Practice Through Educational Approach)
Acronym: CARIATIDE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OEU-ARI-2007/1
Record Dates: First submitted 2008-05-20; First posted 2008-05-21 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2011-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; hormone therapy; aromatase inhibitor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Standard therapy
- 2: Standard therapy + educational material

SUMMARY:
This observational study is restricted to postmenopausal women with hormone-sensitive early breast cancer, who have decided to take prescribed adjuvant use of AIs, anastrozole or letrozole, according to the current product SmPCs. There is no Investigational Medicinal Product (IMP) to be taken in this observational study. The adjuvant AI medication must not have exceeded thirteen weeks. In CARIATIDE (Compliance of ARomatase Inhibitors AssessmenT In Daily practicE through Educational approach), impact of educational material on women's compliance and persistence rates will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman with hormone sensitive early breast cancer
* Documented decision of treatment with upfront adjuvant AI (either anastrozole or letrozole) according to current SmPC OR current treatment with AI (either anastrozole or letrozole) according to current SmPC, that has not exceeded thirteen weeks

Exclusion Criteria:

* Upfront adjuvant AI medication which has exceeded thirteen weeks at randomisation
* Concomitant adjuvant treatment with tamoxifen or exemestane
* Previous use of adjuvant tamoxifen or exemestane exceeding thirteen weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with hormone sensitive early breast cancer that have been prescribed adjuvant AI medication (aromatase inhibitors; anastrozole or letrozole) according to the current product SmPC. The adjuvant AI medication must not have exceeded thirteen weeks of treatment duration.
Sampling Method: Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The compliance rate for the adjuvant AI medication will be analysed at one year based on the subject's assessment. | once after one year

SECONDARY OUTCOMES:
Persistence rate will be evaluated for the first time after one year and a second time after two years. The Investigator will ask the subject about her persistence as follows: | After one and two years.
Time to treatment discontinuation is defined as number of days between the date of first and last intake of AI medication. Dates for AI treatment start and discontinuation will be documented in the CRF. | After one and two years
Reasons for discontinuation of AI: recurrence, death, physician's recommendation, interactions with other medication, side effects, treatment with other hormone medication than anastrozole or letrozole, unfilled AI prescription, subject's wish, other. | After one and two years

CONTACTS AND LOCATIONS:
Overall Officials: Neven, P. Prof., Principal Investigator — KUL
Locations (164):
- Australia (9):
  - Research Site, Canberra, Australian Capital Territory
  - Research Site, Coffs Harbour, New South Wales
  - Research Site, Newcastle, New South Wales
  - Research Site, Port Macquarie, New South Wales
  - Research Site, Tweed Heads, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, Nambour, Queensland
  - Research Site, Toowoomba, Queensland
  - Research Site, Hobart, Tasmania
- Austria (6):
  - Research Site, Sankt Veit im Jauntal, Carinthia
  - Research Site, Wolfsberg, Carinthia
  - Research Site, Salzburg, Salzburg
  - Research Site, Weiz, Styria
  - Research Site, Linz, Upper Austria
  - Research Site, Vienna, Vienna
- Belgium (27):
  - Research Site, Aalst
  - Research Site, Antwerp
  - Research Site, Arlon
  - Research Site, Bonheiden
  - Research Site, Bornem
  - Research Site, Boussu
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Dendermonde
  - Research Site, Edegem
  - Research Site, Eupen
  - Research Site, Geel
  - Research Site, Geraardsbergen
  - Research Site, Ghent
  - Research Site, Gilly
  - Research Site, Haine-Saint-Paul
  - Research Site, Leuven
  - Research Site, Libramont
  - Research Site, Liège
  - Research Site, Namur
  - Research Site, Ostend
  - Research Site, Ottignies
  - Research Site, Overpelt
  - Research Site, Rocourt
  - Research Site, Seraing
  - Research Site, Tournai
  - Research Site, Turnhout
- Chile (2):
  - Research Site, Temuco, Región de la Araucanía
  - Research Site, Santiago, Santiago Metropolitan
- Colombia (6):
  - Research Site, Medellín, Antioquia
  - Research Site, Barranquilla, Atlántico
  - Research Site, Bogota, Cundinamarca
  - Research Site, Neiva, Huila Department
  - Research Site, Pasto, Nari?o
  - Research Site, Cali, Valle del Cauca Department
- Croatia (3):
  - Research Site, Osijek
  - Research Site, Rijeka
  - Research Site, Zagreb
- Czechia (4):
  - Research Site, Hradec Králové
  - Research Site, Opava
  - Research Site, Ostrava
  - Research Site, Prague
- Finland (2):
  - Research Site, Helsinki
  - Research Site, Tampere
- France (48):
  - Research Site, Alès, Ales
  - Research Site, Annecy, Annecy
  - Research Site, Arpajon, Arpajon
  - Research Site, Beauvais, Beauvais
  - Research Site, Bordeaux, Bordeaux
  - Research Site, Brest, Brest
  - Research Site, Brive-la-Gaillarde, Brive La Gaillarde
  - Research Site, Dechy, Dechy
  - Research Site, Évreux, Evreux
  - Research Site, Grenoble, Grenoble
  - Research Site, Hyères, Hyeres
  - Research Site, Limoges, Limoges
  - Research Site, Lyon, Lyon
  - Research Site, Marseille, Marseille
  - Research Site, Mont-de-Marsan, Mont de Marsan
  - Research Site, Mougins, Mougins
  - Research Site, Nantes, Nantes
  - Research Site, Nice, Nice
  - Research Site, Nîmes, Nimes
  - Research Site, Périgueux, Perigueux
  - Research Site, Perpignan, Perpignan
  - Research Site, Reims, Reims
  - Research Site, Rennes, Rennes
  - Research Site, Rouen, Rouen
  - Research Site, Saint Brieux, Saint Brieux
  - Research Site, Saint-Cyr-sur-Loire, Saint Cyr Sur Loire
  - Research Site, Saint-Grégoire, Saint Gregoire
  - Research Site, Saint-Nazaire, Saint Nazaire
  - Research Site, Toulon, Toulon
  - Research Site, Toulouse, Toulouse
  - Research Site, Valence, Valence
  - Research Site, Villeneuve-sur-Lot, Villeneuve Sur Lot
  - Research Site, Aix-en-Provence
  - Research Site, Avignon
  - Research Site, Colmar
  - Research Site, Créteil
  - Research Site, Cucq
  - Research Site, Gap
  - Research Site, La Seyne-sur-Mer
  - Research Site, Mareuil-lès-Meaux
  - Research Site, Nancy
  - Research Site, Narbonne
  - Research Site, Quimper
  - Research Site, Saint-Jean
  - Research Site, Saint-Mandé
  - Research Site, Strasbourg
  - Research Site, Thonon-les-Bains
  - Research Site, Vannes
- Greece (5):
  - Research Site, Pátrai, Achaia
  - Research Site, Athens, Athens
  - Research Site, Piraeous, Piraeous
  - Research Site, Thessaloniki, Thessaloniki
  - Research Site, Trikala, Trikala
- Italy (6):
  - Research Site, Bologna, Bologna
  - Research Site, Cosenza, Cosenza
  - Research Site, Lido di Camaiore, Lucca
  - Research Site, Pavia, Pavia
  - Research Site, Roma, Roma
  - Research Site, Treviso, Treviso
- Peru (2):
  - Research Site, Lima, Lima Province
  - Research Site, Piura, Piura
- Romania (6):
  - Research Site, Alba Iulia
  - Research Site, Baia Mare
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Oradea
  - Research Site, Suceava
- Sweden (3):
  - Research Site, Karlskrona, Karlskrona
  - Research Site, Skellefte?, Skellefte?
  - Research Site, Stockholm, Stockholm County
- Switzerland (5):
  - Research Site, Baden
  - Research Site, Bern
  - Research Site, Lugano
  - Research Site, Sankt Gallen
  - Research Site, Zurich
- Turkey (Türkiye) (10):
  - Research Site, Ankara
  - Research Site, Diyarbakır
  - Research Site, Eskişehir
  - Research Site, Gaziantep
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kayseri
  - Research Site, Konya
  - Research Site, Malatya
  - Research Site, Mersin
- United Kingdom (18):
  - Research Site, St Albans, Hertfordshire
  - Research Site, Brighton
  - Research Site, Bristol
  - Research Site, Cardiff
  - Research Site, Cheltenham
  - Research Site, Coventry
  - Research Site, Dundee
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Macclesfield
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Nottingham
  - Research Site, Scarborough
  - Research Site, Shrewsbury
  - Research Site, York
- Venezuela (2):
  - Research Site, Valencia, Carabobo
  - Research Site, Caracas, Distrito Federal